CLINICAL TRIAL: NCT05612633
Title: A Phase 2 Open-label Study of Zelavespib (PU-H71) in Subjects With Accelerated Phase Myeloproliferative Neoplasm (AP MPN) or Blast Phase Myeloproliferative Neoplasm
Brief Title: A Study of Zelavespib (PU-H71) in Subjects With AP-MPN or BP-MPN
Acronym: AP-MPN
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Samus Therapeutics Closure
Sponsor: Samus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PU-H71-OS-0204
Record Dates: First submitted 2021-10-04; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Accelerated Phase MPN; Blast Phase MPN
Keywords: myeloproliferative neoplasm
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Intervention Model Description: In Stage 1, up to 2317 subjects will be enrolled and will complete 6 cycles of treatment. If fewer than 2 subjects achieve <CR?/PR?/CBR?/PBR?> in Stage 1, the trial will be stopped for futility. If 2 or more subjects achieve <CR?/PR?/CBR?/PBR?>a response , an additional 33 subjects will be enrolled, enrollment will begin in Stage 2 for a total of 56 subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral zelavespib 100 mg (Other): Oral zelavespib 100 mg will be administered once daily
  Interventions: Drug: zelavespib

INTERVENTIONS:
Drug: zelavespib — Oral zelavespib 100 mg will be administered once daily

SUMMARY:
This is a multicenter, Phase 2 Simon 2-Stage study designed to assess the safety, tolerability, PK, and efficacy of oral zelavespib (PU-H71) administered daily in adults with accelerated phase (10% to 19% blasts in peripheral or bone marrow) myeloproliferative neoplasm, with or without ongoing concomitant treatment with ruxolitinib.

DETAILED DESCRIPTION:
Oral zelavespib 1501050 mg will be administered once daily (QD), in the morning ≥ 1 hour before eating breakfast, for each day of a 21-day cycle, for 6 cycles. Subjects who derive clinical benefit may continue treatment until disease progression, unacceptable toxicity, death, or study termination.

In Stage 1, up to 2317 subjects will be enrolled and will complete 6 cycles of treatment. If fewer than 2 subjects achieve <CR?/PR?/CBR?/PBR?> in Stage 1, the trial will be stopped for futility. If 2 or more subjects achieve <CR?/PR?/CBR?/PBR?>a response , an additional 33 subjects will be enrolled, enrollment will begin in Stage 2 for a total of 56 subjects. . If fewer than 2 subjects achieve a response in Stage 1, the trial will be stopped for futility.

In Cycle 1, subjects will attend 3 clinic visits (Day 1, Day 8, and Day 15) and will be contacted by phone by the site at approximately Day 4 . In subsequent cycles, subjects will attend a clinic visit on Day 1 onlyand will be contacted by phone on Days 8 and 15 so the site staff can inquire about changes in concomitant medications and potential AEs. On days of clinic visits, subjects will arrive at the clinic without eating anything in the morning or taking the study drug. Predose biological samples will be collected for safety laboratory tests and other clinical assessments, and subjects will undergo physical examinations and ECGs. Subjects will receive the study drug at the clinic and at least 1 hour after dosing, breakfast will be provided. On some clinic days, subjects may be required to remain in the clinic for up to 8 hours for additional ECGs and collection of samples for PK testing.

Each subject will participate in the study for approximately 6.5 months , which includes a 28-day screening period, 6 cycles of treatment, and a final follow-up visit 30 days after the final dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide signed informed consent and willing to comply with the requirements and restrictions listed in the informed consent form and in this protocol
2. Aged ≥ 18 years
3. Confirmed diagnosis of accelerated phase (10% to 19% blasts in peripheral blood or bone marrow) MPN arising on the background of previous PMF, PV, or ET
4. Patients taking ruxolitinib must have been taking it for at least 3 months, with a stable dose at least 1 month before Cycle 1 Day 1
5. Eastern Cooperative Oncology Group (ECOG) performance status of 1 to 2
6. Acceptable organ function at screening, defined by the following criteria:

   1. absolute neutrophil count (ANC) ≥ 500/µL
   2. platelet count ≥ 50,000/µL
   3. alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 2 × the upper limit of normal (ULN )
   4. total serum bilirubin ≤ 1.5 × ULN
   5. creatinine clearance > 25 mL/min/1.73 m2 based on the Cockcroft-Gault equation
7. Women of childbearing potential (defined as premenopausal or within 2 years of the onset of menopause, and not surgically sterile) must meet both the following criteria:

   1. negative urine or serum pregnancy test at screening and within 72 hours before the first dose of zelavespib
   2. agree to use one of the following acceptable method of highly effective contraception for the duration of the study and for 13 weeks after the final dose of study treatment
8. Men must agree to the following requirements:

   a. men who are sexually active with women of childbearing potential must agree to the following requirements for the duration of their participation in the study and for 13 weeks after the final dose of study treatment: i. if the method of contraception is abstinence from penile vaginal intercourse as a usual and preferred lifestyle (abstinent on a long-term and persistent basis), men must agree to remain abstinent ii. if having penile vaginal intercourse with a nonpregnant, non-breastfeeding woman of childbearing potential, men must use a male condom, and their female partner must use a highly effective contraceptive method with a failure rate < 1% per year iii. men with a pregnant or breastfeeding partner must agree to remain abstinent from penile vaginal intercourse or use a male condom during each episode of penile penetration iv. men must refrain from donating sperm

Exclusion Criteria:

1. Known active liver disease, including viral hepatitis or cirrhosis
2. Known or suspected infection with human immunodeficiency virus (HIV) or other active infection requiring acute or chronic treatment with systemic antibiotics (conditions requiring topical antibiotics are not exclusionary)
3. Positive for HIV 1 or 2, hepatitis B surface antigen (HBsAg), or anti-hepatitis C virus (HCV) antibodies at screening
4. Previous treatment with a hypomethylating agent
5. Corrected QT interval using Fridericia's formula (QTcF) > 480 ms at screening or baseline ECG based on the median value of ECGs
6. Personal or family history of long QT syndrome or taking any medication within 1 week or 5 half-lives (whichever is longer) before Cycle 1 Day 1 that carries a risk of Torsades de Pointes
7. Left ventricular ejection fraction ≤ 50% or below the institution's lower limit of normal (whichever is lower) by echocardiogram or multigated acquisition (MUGA) scan
8. Coronary artery disease with an ischemic event within 6 months before screening
9. History of a second primary malignancy within 6 months before screening that requires treatment with systemic antineoplastic agents, except for the following, if appropriately treated and considered cured: Stage 1 endometrial cancer, surgically treated cervical or prostate carcinoma, and nonmelanoma skin cancer Note: Subjects who are receiving adjuvant or preventive therapy for indolent cancers may be eligible, and the investigator should discuss with the medical monitor.
10. Any significant uncontrolled medical condition, as determined by the investigator, within 6 months before screening
11. Planned use of antineoplastic agents (chemotherapy or cytotoxic drugs), immunotherapy, experimental therapy, or biologic therapy for treatment of MPN, with the exception of ruxolitinib
12. Use of systemic corticosteroids (ie, prednisone > 20 mg/day or equivalent within 2 weeks before Cycle 1 Day 1
13. Planned or current use of strong cytochrome P450 (CYP)3A4/5, CYP2D6, or CYP2C19 inhibitors or inducers within 1 week or 5 half-lives (whichever is longer, for a maximum of 4 weeks) before Cycle 1 Day 1
14. Planned or current use of herbal preparations/medications within 7 days before Cycle 1 Day 1
15. Previous exposure to zelavespib (PU-H71)
16. Uncontrolled diabetes mellitus, in the opinion of the investigator
17. Any other condition or laboratory abnormality or receiving any other treatment that, in the opinion of the investigator, may increase the risk associated with study participation or that may interfere with interpretation of the study results
18. Active ocular condition (eg, ocular inflammatory disease that, in the opinion of the investigator, may worsen during the course of the study, or a history or anticipation of major ocular surgery (eg, cataract extraction or other intraocular surgery) during the study
19. Currently pregnant or breastfeeding, or planning to become pregnant
20. History of gastrointestinal surgery or current gastrointestinal condition that could affect the absorption of oral medication

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-02-23 (Estimated)

PRIMARY OUTCOMES:
Determine the MTD and safety of PU-H71 in subjects with AP-MPN and BP-MPN | up to 6 months
  Assess the safety profile by measuring Incidence and severity of adverse events (AEs), changes in physical examinations, electrocardiograms (ECGs), vital signs, and clinical laboratory evaluations

IPD SHARING:
Plan to Share IPD: Undecided